CLINICAL TRIAL: NCT03067025
Title: Sleep, Physical Activity and Multiple Sclerosis Symptoms in Pediatric Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Alabama at Birmingham (Other); Queen's University (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Associate Scientist, Research Institute, The Hospital for Sick Children
Other Study IDs: 1000055719
Record Dates: First submitted 2017-01-03; First posted 2017-03-01 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Pediatric Multiple Sclerosis
MeSH Terms: interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 youth with MS
  Interventions: Device: Actigraphy
- 30 healthy control participants
  Interventions: Device: Actigraphy

INTERVENTIONS:
Device: Actigraphy — Actiwatch Spectrum Plus will be worn on the non-dominant wrist 24 hours/day for seven days. Actigraphy is a valid and reliable objective measure of sleep patterns, including sleep quality, duration, and timing when compared to polysomnography (PSG).

SUMMARY:
Most youth with MS experience symptoms such as depression and fatigue. In addition, cognitive issues, especially with attention and memory occur frequently. However, little is known about interventions that might work to improve these symptoms. In other work, the investigators have shown that higher levels of physical activity are associated with lower levels of depression and fatigue. Importantly, sleep problems are frequently encountered in youth with MS, and were seen in 60% of surveyed youth with MS in the investigators preliminary work. Modifiable lifestyle factors such as sleep and physical activity (PA) may play a key role in ameliorating common symptoms in pediatric MS. However, sleep has not been objectively described in pediatric MS, and the relationship between PA and sleep is poorly understood. This study aims to address these gaps.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 10 to 17 years, 11 months;
2. MS diagnosis following standard definitions (IPMSSG);
3. Healthy controls will include any child without a history of disease or disability

Exclusion Criteria:

1. Inability to communicate or understand English;
2. Those within 30 days of a relapse;
3. Children who exhibit severe respiratory problems at baseline (e.g. use of tracheotomy)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There will be a total of 60 participants in this study. The study population consists of both patient participants (pediatric multiple sclerosis patients) and non-patient participants (healthy volunteers).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Sleep quality, duration and timing | 7 days
  This will be determined by actigraphy, using the ActiwatchSpectrum Plus, worn on the non-dominant wrist 24 hours/day for seven days. Participants will also complete a sleep diary, the Children's Behavior Check List Sleep Composite, Children's Sleep Habits Questionnaire (CSHQ) and the Pediatric Sleep Questionnaire to derive contextual information about sleep and to identify sleep problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada